CLINICAL TRIAL: NCT06232447
Title: Effect of Menthol to Non-Menthol Cigarette Switching on Subclinical Inflammatory Biomarkers of Cardiovascular Health: Simulating a Menthol Cigarette Ban
Brief Title: Menthol, Inflammation, and Nicotine Transition Study
Acronym: MINT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rosalind Franklin University of Medicine and Science (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Nancy Jao, Assistant Professor, Rosalind Franklin University of Medicine and Science
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CHP22-366; K01HL164670 (NIH)
Record Dates: First submitted 2024-01-09; First posted 2024-01-30 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Cigarette Smoking; Inflammatory Response
MeSH Terms: conditions — Cigarette Smoking

STUDY DESIGN:
Intervention Model Description: All participants will be asked to switch to smoking non-menthol cigarettes for four weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cigarette Type Switching (Experimental): Participants will be switched from smoking menthol cigarettes to non-menthol cigarettes
  Interventions: Other: Cigarette Type Switching

INTERVENTIONS:
Other: Cigarette Type Switching — Participants will be switched from smoking menthol cigarettes to non-menthol cigarettes for a period of four weeks

SUMMARY:
This study will focus on examining the potential impact of menthol flavoring in cigarettes on biomarkers of systemic inflammation as a subclinical indicator of cardiovascular disease risk.

DETAILED DESCRIPTION:
The goal of this study is to examine how switching from menthol (MC) to non-menthol (NMC) cigarette smoking may impact biomarkers of systemic inflammation, smoking behavior, and subjective responses related to smoking. MC smokers (N=68) will be recruited for a five-week study, with one-week of baseline of MC smoking (Phase 1), followed by four weeks of switching to study-provided, brand-matched NMCs (Phase 2). Biomarkers of systemic inflammation and tobacco exposure will be analyzed from blood samples before, during, and after switching for four weeks (baseline, week 1, week 3, and week 5). Ecological momentary assessment methods will also be gathered to measure patterns of smoking and smoking-related subjective responses (affect, craving).

ELIGIBILITY:
Inclusion criteria

* Men and women between 21-85 years old
* Currently uses menthol cigarettes
* Daily smoking rate of ≥5 cigarettes/day for ≥1 year
* Currently own and regularly use an iOS/Android smartphone device able to download the LifeData application
* Able to read and communicate fluently in English

Exclusion criteria

* Currently pregnant or breastfeeding
* Actively trying to quit smoking
* Current heavy alcohol use
* Frequent use of non-menthol cigarettes, other smoking products, or illicit substances
* History of severe medical/psychiatric condition or treatment

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
high sensitivity C-reactive protein | 4 weeks
  from serum in mg/dL
Fibrinogen | 4 weeks
  from serum in mg/dL
Cytokine Panel 13 | 4 weeks
  from serum in mg/dL

SECONDARY OUTCOMES:
Blood pressure | 4 weeks
  systolic blood pressure and diastolic blood pressure, in mm Hg
Heart rate | 4 weeks
  beats per minute

OTHER OUTCOMES:
Affect | 4 weeks
  Positive and Negative Affect Scale (PANAS)
Urge to smoke | 4 weeks
  Questionnaire on Smoking Urges-Brief (QSU)
Nicotine Dependence | 4 weeks
  Fagerström Test for Cigarette Dependence (FTCD)
Number of cigarettes smoked | 4 weeks
  Self-reported total number of menthol and non-menthol cigarettes smoked per day
CO level | 4 weeks
  in ppm

CONTACTS AND LOCATIONS:
Overall Officials: Nancy C Jao, PhD, Principal Investigator — Rosalind Franklin University of Medicine and Science
Locations (1):
- Rosalind Franklin University of Medicine and Science, North Chicago, Illinois, United States